CLINICAL TRIAL: NCT05246098
Title: REVIVe: Frailty, Rehabilitation, and Outcomes in Critically Ill Adult and Pediatric Survivors of COVID-19 or Acute Respiratory Infection
Brief Title: REVIVe: Frailty, Rehabilitation, and Outcomes in Critically Ill Adult and Pediatric Survivors of COVID-19 or ARI
Acronym: REVIVe
Status: Recruiting | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Critical Care Trials Group (Other)
Responsible Party: Sponsor
Other Study IDs: REVIVe
Record Dates: First submitted 2022-02-15; First posted 2022-02-18 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Respiratory Disease; COVID-19; Viral Infection
MeSH Terms: conditions — Respiration Disorders; COVID-19; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adults: Adult survivors of COVID-19 or acute respiratory infection admitted to participating ICUs. Adults are defined as greater than or equal to, 18 years old. We will include adults with a confirmed diagnosis of COVID-19 or those with suspected or proven acute respiratory infection with onset within 14 days of ICU admission and requiring invasive mechanical ventilation, non-invasive ventilation, or high-flow oxygen therapy.
- Pediatrics: Pediatric survivors of COVID-19, MIS-C, or acute respiratory infection admitted to participating pediatric intensive care units (PICUs). The investigators define children as less than 18 years old. We will include pediatric patients with COVID-19, those with multi-system inflammatory syndrome in children (MIS-C), and those with suspected or proven acute respiratory infection with onset within 14 days of ICU admission and requiring invasive mechanical ventilation, non-invasive ventilation, or high-flow oxygen therapy.

SUMMARY:
Background: Many adults and some children with COVID-19 or acute respiratory infection become critically ill and need advanced life support in the Intensive Care Unit (ICU). Frailty is a medical condition of reduced function and health. Adults with frailty have a lower chance of surviving critical illness. The investigators are still learning about critically ill adults with COVID-19 or acute respiratory infection, and do not have much information on how frailty affects outcomes in critically ill children, with or without COVID-19 or acute respiratory infection. Rehabilitation can help survivors of COVID-19 or acute respiratory infection by improving strength and improve quality of life (QOL).

Objectives: The main goal of this research study is to see if patients with frailty have a lower chance of surviving COVID-19 or acute respiratory infection critical illness and more health problems after survival than patients without frailty. The investigators will also study the types of rehabilitation received by patients with COVID-19 or acute respiratory infection.

Methods: The investigators will include adults and children with COVID-19 or acute respiratory infection who are admitted to the ICUs that participate in the study. The investigators will gather data about each patient, including before and during their illness.

Outcomes: The investigators will collect level of frailty, function, and types of therapy, or rehabilitation received by patients. In adults, the investigators are most interested in learning if frailty influences mortality, or death. In children, the investigators are most interested in whether children with COVID-19 or acute respiratory infection critical illness are more likely to develop frailty. The investigators will also study post-hospital discharge location in survivors (e.g., home, rehabilitation).

Relevance: The COVID-19 pandemic is a global public health crisis. It is critical to understand how COVID-19 and other acute respiratory infection critical illness affects groups of people who are at higher risk, and the impact on outcomes that are important to patients, like functioning and QOL. The results will help policy makers plan post-hospital services for survivors, help healthcare workers understand the importance of rehabilitation practice for patients with COVID-19 or acute respiratory infection, and help researchers develop treatments to improve QOL after COVID-19 or acute respiratory infection.

ELIGIBILITY:
Inclusion Criteria:

* Adult and pediatric survivors of COVID-19 or acute respiratory infection admitted to participating intensive care units (ICUs) and PICUs. The investigators define children as less than, and adults as greater than or equal to, 18 years old, respectively. The investigators will include adults and pediatrics with a confirmed diagnosis of COVID-19, pediatric patients with MIS-C, and adults and pediatrics with suspected or proven acute respiratory infection with onset within 14 days of ICU/PICU admission and requiring invasive mechanical ventilation, non-invasive ventilation, or high flow oxygen therapy.

Exclusion Criteria:

* Patients who were admitted to ICU for <24 hours

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric survivors of COVID-19 or acute respiratory infection admitted to participating intensive care units (ICUs) and PICUs. The investigators define children as less than, and adults as greater than or equal to, 18 years old, respectively. The investigators will include adults and pediatrics with a confirmed diagnosis of COVID-19, pediatric patients with MIS-C, and adults and pediatrics with suspected or proven acute respiratory infection with onset within 14 days of ICU/PICU admission and requiring invasive mechanical ventilation, non-invasive ventilation, or high flow oxygen therapy.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Frailty Score (Adults) | hospital discharge or 6-months post ICU admission, whichever occurs first; 6-months post ICU admission
  Frailty
Functional Status Score (Pediatrics) | hospital discharge or 6-months post ICU admission, whichever occurs first; 6-months post PICU admission
  Frailty (paediatrics)

SECONDARY OUTCOMES:
Katz activities of daily living (ADL; adults) | hospital discharge or 6-months post ICU admission, whichever occurs first; 6-months post ICU admission
  Physical Functional
EQ5D-5L (EuroQoL; Adults) | 6-months post ICU admission
  Physical Functional
COVID-19 Yorkshire Rehab Screen | 6-months post ICU admission
  Physical function; cognition; quality of life; disease symptoms
Pediatric Quality of Life Inventory (PedQL) - Multidimensional Fatigue Scale | 6-months post PICU admission
  Quality of Life; Each item is measured on a 5 point Likert scale with 0 indicating never and 4 indicating almost always.The Likert scores are reversed scored and linearly transform to a 0-100 scale with 0=100, 1-75, 2=50, 3=25, and 4=0. A higher score indicates better health-related quality of life.
Pediatric Quality of Life Inventory (PedQL) - General Well-being Scale | 6-months post PICU admission
  Quality of Life; Each item is measured on a 5 point Likert scale with 0 indicating never and 4 indicating almost always.The Likert scores are reversed scored and linearly transform to a 0-100 scale with 0=100, 1-75, 2=50, 3=25, and 4=0. A higher score indicates better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle E Kho, PT, PhD, Principal Investigator — McMaster University
Locations (28):
- Canada (28):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Sturgeon Community Hopsital, St. Albert, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Children's Hospital of Winnipeg, Winnipeg, Manitoba
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Izaak Walton Killam Hospital for Children, Halifax, Nova Scotia
  - Brantford General Hospital, Brantford, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare Intensive Care Unit, Hamilton, Ontario
  - McMaster Children's Hospital, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Sunnybrook Hospital, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Hôpital Hôtel-Dieu de Lévis, Lévis, Quebec
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - The Centre hospitalier universitaire Sainte-Justine, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
  - Hôpital du Sacré-Cœur de Montréal, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec
  - Hôpital Fleurimont - Sherbrooke, Sherbrooke, Quebec
  - Saskatchewan Health Authority, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No